CLINICAL TRIAL: NCT05509868
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study of PBK_L1704 for the Treatment of Moderate to Severe Acute Pain After Bunionectomy in South Korea
Brief Title: Study of PBK_L1704 for the Treatment of Moderate to Severe Acute Pain After Bunionectomy in South Korea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmbio Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBK_L1704_301
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PBK_L1704 0.35mg (Experimental)
  Interventions: Drug: PBK_L1704 0.35mg
- PBK_L1704 0.5mg (Experimental)
  Interventions: Drug: PBK_L1704 0.5mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PBK_L1704 0.35mg — The subject will receive PBK_L1704 0.35mg/ml by PCA
  Arms: PBK_L1704 0.35mg
Drug: PBK_L1704 0.5mg — The subject will receive PBK_L1704 0.5mg/ml by PCA
  Arms: PBK_L1704 0.5mg
Drug: Placebo — The subject will receive placebo by PCA
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate the analgesic efficacy of PBK_L1704 compared with placebo in patients with moderate to severe acute pain after bunionectomy.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo primary, unilateral, first metatarsal bunionectomy with osteotomy and internal fixation
* Able to understand and comply with the study procedures and requirements, and able to provide written informed consent before any study procedure.

Exclusion Criteria:

* Participated in another oliceridine clinical study.
* Received any investigational drug, device or therapy within 35 days before surgery.
* Clinically significant medical, surgical, postsurgical, psychiatric or substance abuse condition or history of such condition that could confound the interpretation of efficacy, safety or tolerability data in the study.
* American Society of Anesthesiologists (ASA) Physical Status Classification System classification III or worse.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
SPID-48 | 48 hours
  Sum of Pain Intensity Difference over 48 hours (SPID-48), calculated from pain intensity scores measured using the Numeric Rating Scale (NRS; 0-10 points), where 0 indicates no pain and 10 indicates the worst possible pain. SPID-48 represents the time-weighted sum of pain intensity differences from baseline across the 48-hour assessment period. Higher SPID-48 values indicate greater pain relief (better outcome).

SECONDARY OUTCOMES:
Responder rate | 48 hours
  A patient is a responder if their final time-weighted Sum of Pain Intensity Differences from baseline (SPID-48) corresponds to, or is greater than, a 30% improvement.
Time to rescue pain medication use | 48 hours
Proportion of rescue pain medication use | 48 hours
Total rescue pain medication use | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Lee, Principal Investigator — Seoul Asan Medical Center
Locations (1):
- Seoul Asan medical Center, Seoul, South Korea